CLINICAL TRIAL: NCT06594783
Title: Carvedilol Plus Endoscopic Ligation or Not for the Primary Prevention of Esophageal Variceal Bleeding in Carvedilol Non-responders: a Randomized Controlled Trial
Brief Title: Carvedilol Plus EVL or Not for the Primary Prevention of Esophageal Variceal Bleeding in Carvedilol Non-responders
Acronym: CVL-NR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-08-017A
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Esophageal Varices
Keywords: Cirrhosis; Endoscopic variceal ligation; Nonselective beta-blocker; Portal hypertension
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Carvedilol plus EVL group:
  Participants will take carvedilol every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable) and undergo EVL every 3-4 weeks until variceal eradication followed by regular endoscopic follow-up according to the protocol.
  Carvedilol alone group:
  Patients will take carvedilol alone every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol plus endoscopic variceal ligation (Active Comparator): Take carvedilol every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable) and undergo EVL every 3-4 weeks until variceal eradication followed by regular endoscopic follow-up according to the protocol.
  Interventions: Other: Carvedilol plus endoscopic variceal ligation
- Carvedilol alone (Placebo Comparator): Take carvedilol alone every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable).
  Interventions: Drug: Carvedilol alone

INTERVENTIONS:
Other: Carvedilol plus endoscopic variceal ligation — Take carvedilol every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable) and undergo EVL every 3-4 weeks until variceal eradication followed by regular endoscopic follow-up according to the protocol.
  Arms: Carvedilol plus endoscopic variceal ligation
Drug: Carvedilol alone — Take carvedilol alone every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable).
  Arms: Carvedilol alone

SUMMARY:
The goal of this clinical trial is to evaluate whether carvedilol plus endoscopic variceal ligation (EVL) is more effective for the primary prevention of esophageal variceal bleeding than carvedilol alone in carvedilol non-responders. It will also learn about the safety of carvedilol combined with EVL in patients with cirrhosis.

The main questions it aims to answer are:

Whether carvedilol plus EVL is more effective than carvedilol alone in preventing the first esophageal variceal bleeding in cirrhotic patients unresponsive to carvedilol.

What medical problems do participants have when taking carvedilol or taking carvedilol combined with undergoing EVL? Researchers will compare the efficacy and safety of carvedilol with or without EVL in preventing the first esophageal variceal bleeding in cirrhotic patients unresponsive to carvedilol.

Participants will:

Take carvedilol every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable) and undergo EVL every 3-4 weeks until variceal eradication followed by regular endoscopic follow-up according to the protocol, or Take carvedilol alone every day (start from 6.25 mg/d and then titrate to 12.5 mg/d if tolerable).

Visit the clinic once every 2-3 months for checkups and tests. Keep a diary of their vital signs (SBP, DBP, and HR) as well as symptoms.

DETAILED DESCRIPTION:
Gastro-esophageal variceal bleeding is a major complication of portal hypertension and carries a high rate of rebleeding and mortality. How to prevent the first esophageal variceal bleeding (EVB) in patients with cirrhosis and portal hypertension has always been a very important issue. According to the latest Baveno VII consensus on the treatment of portal hypertension published in December 2021, nonselective beta-blockers (NSBB) should be used first to prevent decompensation in patients with clinically significant portal hypertension. Endoscopic variceal ligation (EVL) is recommended for compensated patients with high-risk esophageal varices (EVs) who have contraindications or an intolerance to NSBBs.

Carvedilol is a kind of NSBB and has extra intrinsic anti-α1 adrenergic activity. Carvedilol can reduce hepatic venous pressure gradient (HVPG) better than propranolol, and is currently the drug of choice for the primary prevention of EVB in patients with cirrhosis and CSPH. Although the HVPG-lowering effect of carvedilol is stronger than that of propranolol, up to 38-46% patients with CSPH are still carvedilol non-responders. Follow-up upper gastrointestinal endoscopy of these patients may show EVs become larger, more numerous, or have new red color signs, which indicate the increasing risk of EVB. However, studies discussing treatment options for patients with cirrhosis and EVs who do not respond to carvedilol therapy are scarce.

In this project, the investigators will initiate an open-label randomized controlled trial aiming at comparing the efficacy of carvedilol plus EVL or not for the primary prevention of EVB in cirrhotic patients who are carvedilol non-responders. The investigators will also explore if there is any difference between the two groups in terms of other upper gastrointestinal bleeding, non-bleeding liver decompensation (such as new onset/worsening ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, and hepatorenal syndrome), overall survival, adverse events, tolerability and safety. The investigators will also analyze whether there is a difference of the two groups in preventing the first EVB in patients with varying degrees of cirrhosis who are carvedilol non-responders.

ELIGIBILITY:
Inclusion Criteria:

- Cirrhotic patients with esophageal varices who, after carvedilol treatment, continue to experience variceal enlargement or develop new red color signs.

Exclusion Criteria:

* Age under 18 or over 90 years.
* History of esophageal variceal bleeding.
* Previous treatment for esophageal varices, including endoscopic variceal ligation, endoscopic sclerotherapy, transjugular intrahepatic portosystemic shunt, or surgery.
* Contraindications to non-selective beta-blockers, including severe atrioventricular block, chronic obstructive pulmonary disease (COPD), asthma, uncontrolled diabetes mellitus, or severe peripheral artery disease.
* Presence of end-stage organ diseases, including hepatocellular carcinoma or other terminal cancers, heart failure, or renal failure.
* Pregnant women.
* Refusal to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Esophageal variceal bleeding | 3 years
  The cumulative incidence of esophageal variceal bleeding

SECONDARY OUTCOMES:
Other upper gastrointestinal bleeding | 3 years
  The cumulative incidence of other upper gastrointestinal bleeding
First/further nonbleeding liver decompensation | 3 years
  Events that defined first/further nonbleeding liver decompensation were based on the Baveno VII consensus.
Overall survival | 3 years
Adverse events | 3 years

OTHER OUTCOMES:
Primary and secondary outcomes categorized by Child-Pugh class in the subgroup analysis | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung CS, Chang PF, Liao CH, Lee TH, Chen Y, Lee YC, Wu MS, Wang HP, Ni YH. Differences of microbiota in small bowel and faeces between irritable bowel syndrome patients and healthy subjects. Scand J Gastroenterol. 2016;51(4):410-9. doi: 10.3109/00365521.2015.1116107. Epub 2015 Nov 23. PMID 26595305
- [Background] Fernandez M, Semela D, Bruix J, Colle I, Pinzani M, Bosch J. Angiogenesis in liver disease. J Hepatol. 2009 Mar;50(3):604-20. doi: 10.1016/j.jhep.2008.12.011. Epub 2008 Dec 31. PMID 19157625
- [Background] Fernandez M, Vizzutti F, Garcia-Pagan JC, Rodes J, Bosch J. Anti-VEGF receptor-2 monoclonal antibody prevents portal-systemic collateral vessel formation in portal hypertensive mice. Gastroenterology. 2004 Mar;126(3):886-94. doi: 10.1053/j.gastro.2003.12.012. PMID 14988842
- [Background] Schubert K, Olde Damink SWM, von Bergen M, Schaap FG. Interactions between bile salts, gut microbiota, and hepatic innate immunity. Immunol Rev. 2017 Sep;279(1):23-35. doi: 10.1111/imr.12579. PMID 28856736
- [Background] Wahlstrom A, Sayin SI, Marschall HU, Backhed F. Intestinal Crosstalk between Bile Acids and Microbiota and Its Impact on Host Metabolism. Cell Metab. 2016 Jul 12;24(1):41-50. doi: 10.1016/j.cmet.2016.05.005. Epub 2016 Jun 16. PMID 27320064
- [Background] Ridlon JM, Alves JM, Hylemon PB, Bajaj JS. Cirrhosis, bile acids and gut microbiota: unraveling a complex relationship. Gut Microbes. 2013 Sep-Oct;4(5):382-7. doi: 10.4161/gmic.25723. Epub 2013 Jul 12. PMID 23851335
- [Background] Wiest R, Lawson M, Geuking M. Pathological bacterial translocation in liver cirrhosis. J Hepatol. 2014 Jan;60(1):197-209. doi: 10.1016/j.jhep.2013.07.044. Epub 2013 Aug 28. No abstract available. PMID 23993913
- [Background] Baffy G. Potential mechanisms linking gut microbiota and portal hypertension. Liver Int. 2019 Apr;39(4):598-609. doi: 10.1111/liv.13986. Epub 2018 Nov 9. PMID 30312513
- [Background] Arab JP, Martin-Mateos RM, Shah VH. Gut-liver axis, cirrhosis and portal hypertension: the chicken and the egg. Hepatol Int. 2018 Feb;12(Suppl 1):24-33. doi: 10.1007/s12072-017-9798-x. Epub 2017 May 26. PMID 28550391
- [Background] Pande A, Kumar Sarin S, Jindal A, et al. Efficacy of carvedilol, endoscopic variceal ligation (EVL) or a combination for the prevention of first variceal bleed in child B and C cirrhosis with high risk varices: a randomized controlled trial. Hepatology 2019;v70:96A
- [Background] Giuffre M, Dupont J, Visintin A, Masutti F, Monica F, You K, Shung DL, Croce LS; NSBB-Elasto-Response-Prediction Group. Predicting response to non-selective beta-blockers with liver-spleen stiffness and heart rate in patients with liver cirrhosis and high-risk varices. Hepatol Int. 2025 Apr;19(2):460-471. doi: 10.1007/s12072-024-10649-7. Epub 2024 Apr 25. PMID 38664292
- [Background] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Background] Wani ZA, Mohapatra S, Khan AA, Mohapatra A, Yatoo GN. Addition of simvastatin to carvedilol non responders: A new pharmacological therapy for treatment of portal hypertension. World J Hepatol. 2017 Feb 18;9(5):270-277. doi: 10.4254/wjh.v9.i5.270. PMID 28261384
- [Background] Merkel C, Bolognesi M, Sacerdoti D, Bombonato G, Bellini B, Bighin R, Gatta A. The hemodynamic response to medical treatment of portal hypertension as a predictor of clinical effectiveness in the primary prophylaxis of variceal bleeding in cirrhosis. Hepatology. 2000 Nov;32(5):930-4. doi: 10.1053/jhep.2000.19322. PMID 11050041
- [Background] Jachs M, Hartl L, Simbrunner B, Bauer D, Paternostro R, Balcar L, Hofer B, Pfisterer N, Schwarz M, Scheiner B, Stattermayer AF, Pinter M, Trauner M, Mandorfer M, Reiberger T. Carvedilol Achieves Higher Hemodynamic Response and Lower Rebleeding Rates Than Propranolol in Secondary Prophylaxis. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2318-2326.e7. doi: 10.1016/j.cgh.2022.06.007. Epub 2022 Jul 14. PMID 35842118
- [Background] Reiberger T, Ulbrich G, Ferlitsch A, Payer BA, Schwabl P, Pinter M, Heinisch BB, Trauner M, Kramer L, Peck-Radosavljevic M; Vienna Hepatic Hemodynamic Lab. Carvedilol for primary prophylaxis of variceal bleeding in cirrhotic patients with haemodynamic non-response to propranolol. Gut. 2013 Nov;62(11):1634-41. doi: 10.1136/gutjnl-2012-304038. Epub 2012 Dec 18. PMID 23250049
- [Background] Kaplan DE, Ripoll C, Thiele M, Fortune BE, Simonetto DA, Garcia-Tsao G, Bosch J. AASLD Practice Guidance on risk stratification and management of portal hypertension and varices in cirrhosis. Hepatology. 2024 May 1;79(5):1180-1211. doi: 10.1097/HEP.0000000000000647. Epub 2023 Oct 23. No abstract available. PMID 37870298
- [Background] Banares R, Moitinho E, Matilla A, Garcia-Pagan JC, Lampreave JL, Piera C, Abraldes JG, De Diego A, Albillos A, Bosch J. Randomized comparison of long-term carvedilol and propranolol administration in the treatment of portal hypertension in cirrhosis. Hepatology. 2002 Dec;36(6):1367-73. doi: 10.1053/jhep.2002.36947. PMID 12447861
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Sharma M, Singh S, Desai V, Shah VH, Kamath PS, Murad MH, Simonetto DA. Comparison of Therapies for Primary Prevention of Esophageal Variceal Bleeding: A Systematic Review and Network Meta-analysis. Hepatology. 2019 Apr;69(4):1657-1675. doi: 10.1002/hep.30220. Epub 2019 Feb 20. PMID 30125369
- [Background] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2019 Apr 20;393(10181):1597-1608. doi: 10.1016/S0140-6736(18)31875-0. Epub 2019 Mar 22. PMID 30910320
- [Background] Gluud LL, Krag A. Banding ligation versus beta-blockers for primary prevention in oesophageal varices in adults. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD004544. doi: 10.1002/14651858.CD004544.pub2. PMID 22895942
- [Background] Sarin SK, Lamba GS, Kumar M, Misra A, Murthy NS. Comparison of endoscopic ligation and propranolol for the primary prevention of variceal bleeding. N Engl J Med. 1999 Apr 1;340(13):988-93. doi: 10.1056/NEJM199904013401302. PMID 10099140
- [Background] Garcia-Tsao G, Lim JK; Members of Veterans Affairs Hepatitis C Resource Center Program. Management and treatment of patients with cirrhosis and portal hypertension: recommendations from the Department of Veterans Affairs Hepatitis C Resource Center Program and the National Hepatitis C Program. Am J Gastroenterol. 2009 Jul;104(7):1802-29. doi: 10.1038/ajg.2009.191. Epub 2009 May 19. PMID 19455106
- [Background] El-Serag HB, Everhart JE. Improved survival after variceal hemorrhage over an 11-year period in the Department of Veterans Affairs. Am J Gastroenterol. 2000 Dec;95(12):3566-73. doi: 10.1111/j.1572-0241.2000.03376.x. PMID 11151893
- [Background] Sanyal AJ, Bosch J, Blei A, Arroyo V. Portal hypertension and its complications. Gastroenterology. 2008 May;134(6):1715-28. doi: 10.1053/j.gastro.2008.03.007. No abstract available. PMID 18471549